

Title: AZILECT Tablets Special Drug Use-Results Survey "Survey on Long-term Safety"

NCT Number: NCT03727139

Statistical analysis plan Approve Date: 15-Apr-2022

Certain information within this statistical analysis plan has been redacted (ie, specific content is masked irreversibly from view with a black/blue bar) to protect either personally identifiable information or company confidential information.

This may include, but is not limited to, redaction of the following:

- Named persons or organizations associated with the study.
- Patient identifiers within the text, tables, or figures or in by-patient data listings.
- Proprietary information, such as scales or coding systems, which are considered confidential information under prior agreements with license holder.
- Other information as needed to protect confidentiality of Takeda or partners, personal information, or to otherwise protect the integrity of the clinical study.

If needed, certain appendices that contain a large volume of personally identifiable information or company confidential information may be removed in their entirety if it is considered that they do not add substantially to the interpretation of the data (eg, appendix of investigator's curriculum vitae).

Note; This document was translated into English as the language on original version was Japanese.

# The and subject to the applicable Terms of Use applica Statistical Analysis Plan

Name of product

Survey title

Protocol Number

Survey Sponsor

Takeda Pharmaceutical Company Limited Property of Lakeda. Director of Biostatistics Department

Seal

Month Day, Year

#### Table of Contents

| L | ist of | Tern | ns and Abbreviations | 4 |
|---|---|---|---|---|
| A | nalys | sis Po | opulations | 6 |
| S | afety | Spec | rification (Important Identified Risks, Important Potential Risks, and Important | |
| | Mis | ssing | Information) | 7 |
| Η | andli | ng of | f Time Windows | 8 |
| 1 | Nuı | mber | of survey sites, number of patients enrolled, and disposition of patients | 9 |
| | 1 1 | Dis | nosition of natients (Patient disposition diagram) | و د |
| 2 | Patient background | | | . 11 |
| | 2.1 | Pati | ient background | . 11 |
| 3 | Tre | atme | nt details | . 13 |
| | 3.1 | Det | tailed use of this drug | .13 |
| | 3.2 | Stat | tus of treatment compliance with this drug | .13 |
| | 3.3 | Det | ailed use of levodopa | .13 |
| | 3.4 | Det | tailed use of drugs to treat Parkinson's disease other than this drug and levodopa | . 14 |
| | 3.5 | Det | tailed use of concomitant drugs (Parkinson's disease medication) | . 14 |
| | 3.6 | Det | tailed use of concomitant drugs (other than drugs to treat Parkinson's disease) | . 14 |
| | 3.7 | | | |
| | | dis | sease | . 14 |
| | | | tribution of dose by age and body weight | |
| 4 | | - | ata | |
| | 4.1 | Inci | idence of adverse events and adverse drug reactions/infections | |
| | 4 | .1.1 | Incidence of adverse events | .16 |
| | 4 | .1.2 | Incidence of adverse drug reactions/infections | .16 |
| | 4 | .1.3 | Incidence of adverse events and adverse drug reactions/infections relevant to the | |
| | | | safety specification | .17 |
| | 4 | - 1 | Average event duration per day of adverse drug reactions/infections relevant to the | |
| | • | \'/ F | safety specification | .22 |
| | 4.2 | Inci | idence of adverse events and adverse drug reactions/infections in patients excluded | |
| 9 | 3/- | fro | om the safety analysis population | .22 |
| | 4 | .2.1 | Incidence of adverse events in patients excluded from the safety analysis population. | .22 |
| | 4 | .2.2 | | |
| | | | analysis population | .23 |
| | 4.3 | Inci | idence of adverse events and adverse drug reactions/infections by seriousness, time to | |
| | | on | nset, outcome, and causal relationship to this drug. | .23 |

| 4.3.1 Incidence of adverse events by seriousness, time to onset, outcome, and causal | |
|---|---|
| relationship to this drug | 23 |
| 4.3.2 Incidence of adverse drug reactions/infections by seriousness, time to onset, and | 24<br>26 of USE |
| outcome | 24 |
| 4.4 Factors likely affecting the safety | 26 |
| 4.4.1 Incidence of adverse drug reactions/infections by patient background and treatment | "M" |
| factor | 26 |
| 4.4.2 Incidence of adverse drug reactions/infections by sex | * |
| 4.4.3 Incidence of adverse drug reactions/infections by age category (1) | 28 |
| 4.4.4 Incidence of adverse drug reactions/infections by age category (2) | 28 |
| 4.4.5 Incidence of adverse drug reactions/infections by duration of Parkinson's disease | |
| 4.4.6 Incidence of adverse drug reactions/infections by presence or absence of concurrent | |
| diseases | 30 |
| 4.4.7 Incidence of adverse drug reactions/infections by body weight | 30 |
| 4.4.8 Incidence of adverse drug reactions/infections by presence or absence of concurrent | |
| renal disorder | 30 |
| 4.4.9 Incidence of adverse drug reactions/infections by presence or absence of concurrent | |
| hepatic disorder | 30 |
| 4.4.10 Incidence of adverse drug reactions/infections by treatment stage | 31 |
| 4.4.11 Incidence of adverse drug reactions/infections by daily dose | 31 |
| 4.4.12 Incidence of adverse drug reactions/infections by presence or absence of dementia | 31 |
| 4.4.13 Incidence of adverse drug reactions/infections by presence or absence of dyskinesia | |
| 5 Efficacy data | 33 |
| 5.1 UPDRS Part III total score over time | 33 |
| 5.2 UPDRS Part III tremor score over time | |
| 5.3 UPDRS Part III akinesia/hypokinesia score over time | 33 |
| 5.4 UPDRS Part III rigidity score over time | 33 |
| 5.5 Factors likely affecting the efficacy | 34 |
| 5.54 Factors likely affecting the efficacy | 34 |
| 5.5.2 UPDRS Part III total score by age category and number of concomitant drugs | 35 |
| 5.5.3 Number of patients continuing treatment with this drug by age category and number | |
| of concomitant drugs | 35 |
| 5.5.4 Number of patients continuing treatment with this drug by age category | 35 |
| 5.5.1 Factors likely affecting the efficacy | 36 |
| 6 Incidence of adverse drug reactions/infections in the additional pharmacovigilance plan | 37 |
| 6.1 Incidence of adverse drug reactions/infections in the additional pharmacovigilance plan | |
| (Attached Form 12) | 37 |

| 7.1 Su | ammary of patients in the | e post-marketing survey/stud | ly (Attached Form 16) | 38 |
|---|---|---|---|---|
| History of | this document (Version of | control) | | 39 |
| | | | | Ó |
| | | | | -KINS |
| | | | | √ <sub>©</sub> , |
| | | | | 3016 |
| | | | | lice |
| | | | 3 | • |
| | | | *0 | |
| | | | . 00 | |
| | | t-marketing survey/study e post-marketing survey/study control) | SUDI | |
| | | by | | |
| | | 4 | | |
| | | e O | | |
| | | 11/5 | | |
| | C | KCio | | |
| | nin's | | | |
| | 7.CO1 | | | |
| | " KOII. | | | |
| | 401 | | | |
| 93 | * | | | |
| 19Ke | | | | |
| ,01 | | | | |
| eka | | | | |
| Υ | | | | |

#### List of Terms and Abbreviations

- This drug: AZILECT Tablets is abbreviated as "this drug".
- Adverse events: Adverse events that occurred after administration of this drug
- ADRs: Adverse drug reactions/infections, defined as adverse events other than those assessed as causally "not related" to this drug by the survey physician. This statistical analysis plan uses "adverse drug reactions/infections" in titles and ADRs in main text and table columns.
- Serious adverse event: An adverse event assessed as "serious" by the survey physician. Also, events listed in the MedDRA Code List (PT code) of the Important Medical Events List are handled as serious events, even if the event is assessed as "non-serious" by the survey physician.
- "Related" to this drug: Adverse events with a causal relationship to this drug other than "not related" are handled as "related", and adverse events with a causal relationship to this drug of "not related" are handled as "not related".
- Summary statistics: This includes the number of patients, mean, standard deviation, maximum, minimum, and quartiles.
- Number of days after administration: The day before initiation of treatment is counted as −1 day,
   and the day of initiation of treatment is counted as 1 day.
- Treatment duration (days): Therapy end date Therapy start date + 1
- Disease duration (years): Calculated as (Date of first administration of this drug Date of disease onset + 1)/365.25. If the month and day of disease onset are unknown, January 1 shall be used. If the day of disease onset is unknown, 1 shall be used as the day. The calculated value shall be rounded to the first decimal place.
- Patients without collected CRFs: Patients who were enrolled but whose CRFs were not collected
- Patients with collected CRFs: Patients who were enrolled and whose CRFs were collected
- Time to adverse event (or ADR) onset: Calculated as "Date of onset of the adverse event (or ADR) – Date of first administration of this drug + 1".
  - If the month and day of onset of the adverse event (or ADR) are unknown, January 1 shall be used in the calculation. However, if the year of first administration of this drug is the same as the year of onset of the adverse event (or ADR), the month and day of first administration of this drug shall be used in the calculation.
  - If the day of onset of the adverse event (or ADR) is unknown, 1 shall be used as the day. However, if the year and month of first administration of this drug are the same as the year

and month of onset of the adverse event (or ADR), the day of first administration of this drug shall be used in the calculation.

- Unified Parkinson's Disease Rating Scale (UPDRS) Part III total score: Calculated by summing the following scores: "Speech", "Facial expression", "Resting tremor (face, left hand, right hand, left foot, right foot)", "Hand kinetic tremor or postural tremor (left, right)", "Rigidity (neck, left upper extremity, right upper extremity, left lower extremity, right lower extremity)", "Finger tapping (left, right)", "Hand movements (left, right)", "Pronation-supination movements of hands (left, right)", "Leg agility (left, right)", "Arising from chair", "Posture", "Gait", "Postural stability", "Bradykinesia and hypokinesia".
   Unified Parkinson's Disease Rating Scale (UPDRS) Part III
- Unified Parkinson's Disease Rating Scale (UPDRS) Part III tremor score: Calculated by summing
  the following scores: "Resting tremor (face, left hand, right hand, left foot, right foot)" and "Hand
  kinetic tremor or postural tremor (left, right)".
- Unified Parkinson's Disease Rating Scale (UPDRS) Part III akinesia/hypokinesia score:
   Calculated by summing the following scores: "Finger tapping (left, right)", "Hand movements (left, right)", "Pronation-supination movements of hands (left, right)", "Leg agility (left, right)", and "Bradykinesia and hypokinesia".
- Unified Parkinson's Disease Rating Scale (UPDRS) Part III rigidity score: Calculated by summing the following scores: "Rigidity (neck left upper extremity, right upper extremity, left lower extremity, right lower extremity)".

   The part of the part o

#### **Analysis Populations**

The analysis populations of "safety analysis population" and "efficacy analysis population" will be

population is defined as the patients who received this drug, had no major protocol violations, and were evaluable for safety. More specifically, the safety analysis population will exclude patients meeting the following conditions, among those with the CRF data locked:

No administration of this drug

Administration of this drug Enrollment outside the enrollment period

Enrollment 15 days or more after the date of prescription of this drug

Prescription of this drug outside of the contract period

No information on presence or absence of adverse events

Withdrawal of consent

Efficacy and

#### • Efficacy analysis population

and subject This population is defined as a subset of the patients in the safety analysis population who had no major protocol violations and were evaluable for efficacy. More specifically, the efficacy analysis population will exclude patients meeting the following conditions,

- · No target disease
- Property of Fakedai. For non-comm No target disease
   Administration of contraindicated medication for this drug (Parkinson's disease medication)

#### Safety Specification (Important Identified Risks, Important Potential Risks, and Important **Missing Information**)

- Important identified risks
- of "(4)1

  y of "(4)1

  Frogeth of Takeda. For non-commercial use only and subject to a subject to Dyskinesia: Events falling under the adverse event category of "(4) Dyskinesia" in the

#### **Handling of Time Windows**

For observation items, data that are evaluable (i.e., not missing and determined to be included in analysis) shall be handled in accordance with the following.

The data that are evaluable and within the allowable time window shall be used. If there are multiple evaluable data within the same allowable time window, the one closest to the standard implementation time point of the examination, observation, or assessment shall be used. If the magnitude of difference from the standard implementation time point is the same, or if the standard implementation time point is not specified, the later data shall be used. The magnitude of the difference from the standard implementation time point shall be determined based on the number of days after administration.

Unified Parkinson's Disease Rating Scale (UPDRS) Part III

| Unified Parkinson's Disease Rating Scale (UI | DKS) Falt III | |
|---|---|---|
| Time point of assessment | Standard implementation time point | Allowable time window Number of days after administration |
| At initiation of treatment with this drug (Baseline) | Number of days<br>after<br>administrat<br>ion: | -30 - 1 |
| At 6 months of treatment | Number of days after administrat ion: | 2 - 273 |
| At 12 months of treatment | Number of days<br>after<br>administrat<br>ion: | 274 - 456 |
| At 18 months of treatment | Number of days<br>after<br>administrat<br>ion: | 457 - 638 |
| At 24 months of treatment or discontinuation | Number of days<br>after<br>administrat<br>ion: | 639 - 821 |
| Final assessment | Number of days<br>after<br>administrat<br>ion: | 2 - 821 |

#### 1 Number of survey sites, number of patients enrolled, and disposition of patients

#### 1.1 Disposition of patients (Patient disposition diagram)

Analysis set: All enrolled patients (Enrolled patients)

Analysis item(s): Enrolled patients

Number of survey sites

Patients without collected CRFs
Patients with collected CRFs
Patients excluded from the
safety analysis population\*

Reasons for exclusion

(patients counted under all

applicable categories)

[No administration of this drug,

Administration of this drug before the contractual period, Enrollment outside the enrollment period, Enrollment 15 days or more after the date of prescription of this drug, Prescription of this drug outside of the contract period, No information on presence or absence of adverse events,

icable Terms of Use

Withdrawal of consent]

Safety analysis population
Patients excluded from the
efficacy analysis population\*

Reasons for exclusion (patients counted under all applicable categories)

Efficacy analysis population

[No target disease, Administration of contraindicated medication for this drug (Parkinson's disease medication)]

Analyses of the above items will be performed as follows, and a patient disposition diagram will be constructed.

For enrolled patients, the number of survey sites shall also be presented. The same medical institution with different departments in the survey shall be counted as one medical institution. Reasons for exclusion are broken into categories; if there are no patients in a certain category, "0" will be indicated. For patients excluded from the safety or efficacy analysis population, the numbers of patients will be counted by reason for exclusion, and a tabulated list will be prepared.

\*Patients excluded from the safety analysis population refer to patients whose CRF data locked and who were excluded from the safety analysis population. Patients excluded from the efficacy analysis population refer to patients who

Analytical methods:

were in the safety analysis population and who were excluded from the efficacy

Property of Takeda: For non-commercial use only and subject to the applicable Tames of use

#### 2 Patient background

#### Patient background 2.1

Analysis set: Safety analysis population

Analysis item(s):

80, 80<= - <-Max]

[0<= - <5, 5<= - <10, 10<= - <15, 15<= - <-Max, Unknown]

[Outpatient, Inpatient] Age (years)

Duration of Parkinson's disease

(years)

Inpatient/outpatient status (at

initiation of treatment with this

drug)

Concurrent diseases [No, Yes]

Specific concurrent diseases

[Diabetes mellitus, Hypertension, (patients counted under all

applicable categories) Dyslipidemia, Hyperuricaemia]

[Hepatic steatosis, Alcoholic hepatitis, Lifestyle-related disease

Chronic hepatitis, Hepatic cirrhosis]

Nephrotic syndrome, Glomerulonephritis, Hepatic disease

Chronic renal failure]

Renal disease [Dementia, Pneumonia aspiration,

Constipation]

Other diseases

Dementia [No, Yes]

Height (cm) Min < = < = 140,141 < = < = 150,151 < = <

=160,161 < = - < =170,171 < = - < = Max, Not

measured].

[Min < = < 50,50 < = < 65,65 < = < = Max,Body weight (kg)

Not measured].

Smoking history [Never smoker, Current smoker, Former

smoker, Unknown]

Modified Hoehn & Yahr [0, 1, 1.5, 2, 2.5, 3, 4, 5]

Property of Takedai. For Po Severity scale (Stage)

Levodopa use at initiation of [No, Yes]

treatment with this drug

Wearing-off phenomenon [No, Yes] Note: Only in patients given levodopa at initiation of treatment with this drug

Dyskinesia

[No, Yes]

Note: Only in patients given levodopa at initiation of treatment with this drug

UPDRS Part III total score (at initiation of treatment with this

drug)

Tremor score (at initiation of treatment with this drug)

Akinesia/hypokinesia score (at initiation of treatment with this

drug)

Rigidity score (at initiation of treatment with this drug)

Treatment stage

[Min<= - <=10, 11<= - <=20, 21<= - <=30, 1 [1VIII] = - <=10, 11<= - <=20, 21<= - <=3
31<= - <=40, 41<= - <=50, 51<= - <=60,
61<= - <=Max]

[Δ7II FCT alone: Δ7II FCT + other

[AZILECT alone; AZILECT + other Parkinson's disease m. ' Parkinson's disease medication; Combined anout wearing-o

...on; Combined with levodopa
other Parkinson's disease medication, w
wearing-off phenomenon; Combined win
levodopa, with wearing-off phenomenon
For the above analysis items, discrete data will be summarized using frequen
tabulation and continuous data will be summarized using summary statistics. with only levodopa, without wearing-off
phenomenon; Combined with levodopa and
other Parkinson's disease medication, without
wearing-off phenomenon; Combined with
levodopa, with wearing-off phenomenon]
For the above analysis items, discrete data will be summarized using frequency other Parkinson's disease medication, without

12

#### 3 Treatment details

#### 3.1 Detailed use of this drug

Analysis set: Safety analysis population

Analysis item(s): Daily dose [1 mg, 0.5 mg, Other]

Overdose [No, Yes]

Any adverse event due to overdose [No, Yes]

Reason for use (at initial dose) [Because of the patient's mild hepatic

Note: Only when the daily dose was impairment, low body weight, advanced

"0.5 mg" age, or concurrent CYP1A2 inhibitor

use; Other]

Treatment duration (months) [0 <= - <= 6, 7 <= - <= 12, 13 <= - <= 18,

19<= - <= Max]

Reason for treatment discontinuation [Achievement of treatment goal;

Adverse event onset; No return to survey

site (including referral to another

hospital); Pregnancy; Inadequate

effectiveness; Withdrawal of consent;

Other]

Analytical For the above analysis items, discrete data will be summarized using frequency

methods: tabulation and continuous data will be summarized using summary statistics.

#### 3.2 Status of treatment compliance with this drug

Analysis set: Safety analysis population

Analysis item(s): Status of treatment [90% or more, 70% or more, 50% or more, <50%,

compliance with this drug No doses were taken, or treatment compliance was

unknown]

Analytical For the above analysis item, data will be summarized using frequency tabulation

methods: by time point of assessment (i.e., at 6 months, 12 months, 18 months, and 24

months of treatment or discontinuation).

#### 3.3 Detailed use of levodopa

Analysis set: Safety analysis population

Analysis item(s): Levodopa use [No, Yes]

Daily dose [<200 mg, 200 to <400 mg, ≥400 mg]

Treatment duration (months) [0<= - <=6, 7<= - <=12, 13<= - <=18,

 $19 \le - \le Max$ 

Analytical For the above analysis items, discrete data will be summarized using frequency

methods: tabulation and continuous data will be summarized using summary statistics.

#### 3.4 Detailed use of drugs to treat Parkinson's disease other than this drug and levodopa

Analysis set: Safety analysis population

Analysis item(s): Any drugs to treat Parkinson's disease [No, Yes]

other than AZILECT and levodopa

Name of drug

Analytical Frequency tabulation will be performed for the above analysis item.

methods:

#### 3.5 Detailed use of concomitant drugs (Parkinson's disease medication)

Analysis set: Safety analysis population

Analysis item(s): Number of concomitant drugs [0 (AZILECT alone), 1 (AZILECT +

another drug),  $\geq 2$  (AZILECT +  $\geq 2$ 

other drugs)]

Analytical Frequency tabulation will be performed for the above analysis item.

methods:

#### 3.6 Detailed use of concomitant drugs (other than drugs to treat Parkinson's disease)

Analysis set: Safety analysis population

Analysis item(s): Concomitant drugs (Parkinson's disease [No, Yes]

medication)

Analytical Frequency tabulation will be performed for the above analysis item.

methods:

## 3.7 Detailed use of concomitant therapies other than pharmacotherapy for Parkinson's disease

Analysis set: Safety analysis population

Analysis item(s): Use of concomitant medications [No, Yes]

other than medications for

Parkinson's disease

Analytical Frequency tabulation will be performed for the above analysis item.

methods:

#### 3.8 Distribution of dose by age and body weight

Safety analysis population Analysis set:

Analysis item(s): Daily dose

Stratification Age (years)

factor 1:

Stratification Body weight

factor 2:

-<65, 65<= - <75, 75<= - <=Max]

[Min<= - <50, 50<= - <65, 65<= - <=Max]

patients will be stratified first by tion factor 2, with the each strate For the above analysis item, patients will be stratified first by Stratification After the am of Stration of Stration of Stration of Stration of Takeda. For noncommercial use only and subject of Takeda. For noncommercial use only and subject of takeda. Analytical

methods: factor 1 and then by Stratification factor 2, with the discrete data summarized

using frequency tabulation for each stratum of Stratification factor 2.

#### Safety data

#### Incidence of adverse events and adverse drug reactions/infections 4.1

#### 4.1.1 Incidence of adverse events

Analysis set: Safety analysis population

Analysis item(s): Adverse events

Analytical methods: Analyses of the above analysis item will be performed as follows.

- 1. Number of patients with adverse events
- 2. Number of adverse events
- 3. Percentage of patients with adverse events
- 4. Type of adverse events

All analyses will be accounted for as follows.

[Number of patients with adverse events]

Number of patients who experienced adverse events.

[Number of adverse events]

Number of adverse events that occurred. When the same patient experienced multiple episodes of the same adverse event, all episodes will be counted.

[Percentage of patients with adverse events]

Calculated as "Number of patients with adverse events/Number of patients in the safety analysis population x 100"

[Type of adverse events]

- Adverse events will be coded using MedDRA/J. Events will be classified by SOC and then tabulated by PT. If the SOC is "Investigations", events will be sorted by HLGT (in ascending order of HLGT code, without output) and then tabulated by PT.
- The SOCs will be listed in the internationally agreed order for presentation of the number and percentage of patients with adverse events. When the same patient experienced multiple episodes of the same SOC, they will be counted only once for the SOC.
- The PTs will be listed in ascending order of PT code for presentation of the number and percentage of patients with adverse events. When the same patient experienced multiple episodes of the same PT, they will be counted only once for the PT.

# Property of Takedai. For non-ch 4.1.2 Incidence of adverse drug reactions/infections

Safety analysis population Analysis set:

**ADRs** Analysis item(s):

Analytical methods:

Analyses of the above analysis item will be performed as follows.

- 1. Number of patients with ADRs
- 2. Number of ADRs
- 3. Percentage of patients with ADRs
- 4. Type of ADRs

All analyses will be accounted for as follows.

[Number of patients with ADRs]

• Number of patients who experienced ADRs.

#### [Number of ADRs]

 Number of ADRs When the same patient experienced multiple episodes of the same ADR, all episodes will be counted.

[Percentage of patients with ADRs]

 Calculated as "Number of patients with ADRs/Number of patients in the safety analysis population x 100"

#### [Type of ADRs]

- ADRs will be coded using MedDRA/J. Events will be classified by SOC and then tabulated by PT. If the SOC is "Investigations", events will be sorted by HLGT (in ascending order of HLGT code, without output) and then tabulated by PT.
- The SOCs will be listed in the internationally agreed order for
  presentation of the number and percentage of patients with ADRs.
  When the same patient experienced multiple episodes of the same
  SOC, they will be counted only once for the SOC.
- The PTs will be listed in ascending order of PT code for presentation of the number and percentage of patients with ADRs. When the same patient experienced multiple episodes of the same PT, they will be counted only once for the PT.

# 4.1.3 Incidence of adverse events and adverse drug reactions/infections relevant to the safety specification

# 4.1.3.1 Incidence of adverse events relevant to the safety specification (Tabulation by risk item)

Analysis set: Safety analysis population

Analysis item(s): Adverse events relevant to the important identified risks in the safety

specification (i.e., Orthostatic hypotension, Somnolence and sudden onset

of sleep, Psychiatric symptoms such as hallucinations, Dyskinesia)

Stratification factors: Total

Seriousness [Serious, Non-serious]

Time to onset (days)  $[1 \le -1 \le 27, 28 \le -1 \le 55, 56 \le -1]$ 

<=83, 84<= - <=167, 168<= -

<=251, 252<= - <=365, 366<= -

 $\leq = Max$ 

Outcome [Resolved, Resolving, Not

resolved, Resolved with sequelae,

Death (from the event), Unknown]

[Related, Not related]

[Mild, Moderate, Severe]

Causal relationship to this drug

Severity (Somnolence and sudden

onset of sleep, Psychiatric

symptoms such as hallucination,

Dyskinesia)

Fall or trauma (Orthostatic [No, Yes]

hypotension, Psychiatric symptoms such as hallucinations, Dyskinesia)

Accident or injury (Somnolence and [No, Yes]

sudden onset of sleep)

Analytical methods:

Property of Takedai. For non'

For the above analysis item by risk item, the following analysis will be performed for each stratum of stratification factors. For the risk items to be analyzed, the definitions described in the safety specification (important identified risks, important potential risks, and important missing information) shall be followed.

[Number of patients with adverse events]

Number of patients who experienced adverse events.

[Number of adverse events]

 Number of adverse events that occurred. When the same patient experienced multiple episodes of the same adverse event, all episodes will be counted.

[Percentage of patients with adverse events]

• Calculated as "Number of patients with adverse events/Number of patients in the safety analysis population x 100"

[Type of adverse events]

 Adverse events will be coded using MedDRA/J. Events will be classified by SOC and then tabulated by PT. If the SOC is "Investigations", events will be sorted by HLGT (in ascending order of HLGT code, without output) and then tabulated by PT.

- The SOCs will be listed in the internationally agreed order for presentation of the number and percentage of patients with adverse events. When the same patient experienced multiple episodes of the same SOC, they will be counted only once for the SOC. For counting by category, if the episodes fall under different categories of a stratification factor, the episodes will be counted once for each of the categories involved. However, in terms of the stratification factors specified at the end of this section, the episodes will be counted only once in the category of highest priority.
- The PTs will be listed in ascending order of PT code for presentation of the number and percentage of patients with adverse events. When the same patient experienced multiple episodes of the same PT, they will be counted only once for the PT. For counting by category, if the episodes fall under different categories of a stratification factor, the episodes will be counted once for each of the categories involved. However, in terms of the following stratification factors, they will be counted only once in the category of highest priority.

Severity: Severe  $\rightarrow$  Moderate  $\rightarrow$  Mild

Fall or trauma: Yes  $\rightarrow$  No Accident or injury: Yes  $\rightarrow$  No

# 4.1.3.2 Incidence of adverse drug reactions/infections relevant to the safety specification (Tabulation by risk item)

Analysis set: Safety analysis population

Analysis item(s): ADRs relevant to the important identified risks in the safety specification

(i.e., Orthostatic hypotension, Somnolence and sudden onset of sleep,

Psychiatric symptoms such as hallucinations, Dyskinesia)

Stratification factors: Total Serio T'

Seriousness [Serious, Non-serious]

Time to onset (days)  $[1 \le -1 \le 27, 28 \le -1 \le 55, 56 \le -1]$ 

<=83, 84<= - <=167, 168<= -

<=251, 252<= - <=365, 366<= -

 $\leq =Max$ 

Outcome [Resolved, Resolving, Not

resolved, Resolved with sequelae,

Death (from the event), Unknown]

Severity (Somnolence and sudden [Mild, Moderate, Severe] onset of sleep, Psychiatric symptoms such as hallucination, Dyskinesia)

Fall or trauma (Orthostatic [No, Yes]

hypotension, Psychiatric symptoms such as hallucinations, Dyskinesia)

Accident or injury (Somnolence and [No, Yes]

sudden onset of sleep)

Analytical methods:

Cable Terms of Use For the above analysis item by risk item, the following analysis will be performed for each stratum of stratification factors. For the risk items to be analyzed, the definitions described in the safety specification (important identified risks, important potential risks, and important missing information) shall be followed.

[Number of patients with ADRs]

Number of patients who experienced ADRs.

[Number of ADRs]

Number of ADRs When the same patient experienced multiple episodes of the same ADR, all episodes will be counted.

[Percentage of patients with ADRs]

Calculated as "Number of patients with ADRs/Number of patients in the safety analysis population x 100"

#### [Type of ADRs]

- ADRs will be coded using MedDRA/J. Events will be classified by SOC and then tabulated by PT. If the SOC is "Investigations", events will be sorted by HLGT (in ascending order of HLGT code, without output) and then tabulated by PT.
- Property of Takedai. For non-ch The SOCs will be listed in the internationally agreed order for presentation of the number and percentage of patients with ADRs. When the same patient experienced multiple episodes of the same SOC, they will be counted only once for the SOC. For counting by category, if the episodes fall under different categories of a stratification factor, the episodes will be counted once for each of the categories involved. However, in terms of the stratification factors specified at the end of this section, the episodes will be counted only once in the category of highest priority.

The PTs will be listed in ascending order of PT code for presentation of the number and percentage of patients with ADRs. When the same Lategory, if the Lategories of a stratification factor, the Lategories will be counted once for each of the categories involved.

However, in terms of the following stratification factors, they will be counted only once in the category of highest priority.

Severity: Severe 

Moderate 

Mild

Fall or trauma: Yes

Accident or injury: Yes  $\rightarrow$  No

#### Incidence of adverse drug reactions/infections meeting the safety specification by 4.1.3.3 presence or absence of levodopa use (Tabulation by risk item)

Analysis set: Safety analysis population

ADRs relevant to the important identified risks in the safety specification Analysis item(s):

(i.e., Psychiatric symptoms such as hallucinations, Dyskinesia)

Stratification factor 1: Levodopa use [No, Yes]

Stratification factor 2: Total

> Seriousness [Serious, Non-serious]

Time to onset (days) [1<= - <=27, 28<= - <=55, 56<= -

<=83, 84<= - <=167, 168<= -

<=251, 252<= - <=365, 366<= -

 $\leq Max$ 

[Resolved, Resolving, Not

resolved, Resolved with sequelae, Death (from the event), Unknown]

[Mild, Moderate, Severe]

[No, Yes]

Analytical methods: The above analysis item by risk item will be analyzed with stratification

by Stratification factor 1 and Stratification factor 2, in the same manner as

described in Section 4.1.3.2. For the risk items to be analyzed, the

definitions described in the safety specification (important identified risks,

important potential risks, and important missing information) shall be

followed.

### 4.1.4 Average event duration per day of adverse drug reactions/infections relevant to the safety specification

# 4.1.4.1 Average event duration per day of adverse drug reactions/infections relevant to the safety specification (1)

Analysis set: Safety analysis population

Analysis item(s): Average event duration per day (hours)

Analytical methods: For the above analysis item of the ADRs relevant to the important

identified risks in the safety specification (Somnolence, Sudden onset of sleep, Psychiatric symptoms such as hallucination, Dyskinesia), summary statistics (of individual patients' average values) will be calculated for each risk item. For the risk items to be analyzed, the definitions described in the safety specification (important identified risks, important potential

risks, and important missing information) shall be followed.

# 4.1.4.2 Average event duration per day of adverse drug reactions/infections relevant to the safety specification (2)

Analysis set: Safety analysis population

Analysis item(s): Patient ID number

Adverse drug reaction (disease name, disease code)

Average event duration per day (hours)

Severity

Fall or trauma (Psychiatric symptoms such as hallucinations, Dyskinesia)

Accident or injury (Somnolence and sudden onset of sleep)

Analytical methods: For the above analysis item of the ADRs relevant to the important

identified risks in the safety specification (Somnolence, Sudden onset of

sleep, Psychiatric symptoms such as hallucination, Dyskinesia), a

tabulated list will be prepared for each risk item. For the risk items to be

analyzed, the definitions described in the safety specification (important

identified risks, important potential risks, and important missing

information) shall be followed.

# 4.2 Incidence of adverse events and adverse drug reactions/infections in patients excluded from the safety analysis population

#### 4.2.1 Incidence of adverse events in patients excluded from the safety analysis population

Analysis set: Patients excluded from the safety analysis population

Analysis item(s): Adverse events

Analytical methods: The above item will be analyzed in a similar manner to Section 4.1.1.

#### 4.2.2 Incidence of adverse drug reactions/infections in patients excluded from the safety analysis population

Analysis set:

Analysis item(s):

Analytical methods:

- Incidence of adverse events and adverse drug reactions/infections by seriousness, time to onset, outcome, and causal relationship to this drug

  Incidence of adverse events by seriousness, time to onset. Outcome, and causal relationship to this drug

  ysis set: 4.3
- 4.3.1 Incidence of adverse events by seriousness, time to onset, outcome, and causal relationship to this drug

Analysis set: Safety analysis population

Analysis item(s): Adverse events

Stratification factors: Total

> Seriousness [Serious, Non-serious]

Time to onset (days)

<=365, 366 <= - <= Max

Outcome [Resolved, Resolving, Not resolved,

Resolved with sequelae, Death (from the

event), Unknown]

Causal relationship to this [Related, Not related]

For the above analysis item, the following analysis will be performed for Analytical methods: Property of Takedai. For not each stratum of stratification factors.

- Number of patients with adverse events
- 2. Number of adverse events
- 3. Percentage of patients with adverse events
- Type of adverse events

All analyses will be accounted for as follows.

[Number of patients with adverse events]

Number of patients who experienced adverse events.

[Number of adverse events]

Number of adverse events that occurred. When the same patient experienced multiple episodes of the same adverse event, all episodes will be counted.

[Percentage of patients with adverse events]

 Calculated as "Number of patients with adverse events/Number of patients in the safety analysis population x 100"

[Type of adverse events]

- Adverse events will be coded using MedDRA/J. Events will be classified by SOC and then tabulated by PT. If the SOC is "Investigations", events will be sorted by HLGT (in ascending order of HLGT code, without output) and then tabulated by PT.
- The SOCs will be listed in the internationally agreed order for presentation of the number and percentage of patients with adverse events. When the same patient experienced multiple episodes of the same SOC, they will be counted only once for the SOC. For counting by category, episodes in the same SOC will be counted only once in the category of highest priority specified at the end of this section.
- The PTs will be listed in ascending order of PT code for presentation of the number and percentage of patients with adverse events. When the same patient experienced multiple episodes of the same PT, they will be counted only once for the PT. For counting by category, episodes in the same PT will be counted only once in the category of highest priority as shown below.

Seriousness: Serious → Non-serious

Time to onset: 1–27 days  $\rightarrow$  28–55 days  $\rightarrow$  56–83 days  $\rightarrow$  84–167

days  $\rightarrow$  168–251 days  $\rightarrow$  252–365 days  $\rightarrow$  366 days or more

Outcome: Death (from the event)  $\rightarrow$  Resolved with sequelae  $\rightarrow$  Not

resolved  $\rightarrow$  Resolving  $\rightarrow$  Resolved  $\rightarrow$  Unknown

Relationship to this drug: Related → Not related

# 4.3.2 Incidence of adverse drug reactions/infections by seriousness, time to onset, and outcome

Analysis set: Safety analysis population

Analysis item(s): ADRs Stratification factors: Total

Seriousness [Serious, Non-serious]

Time to onset (days)  $[1 \le -1 \le 27, 28 \le -1 \le 55, 56 \le -1 \le 83, 1 \le 10]$ 

84<= - <=167, 168<= - <=251, 252<= -

<=365, 366<= - <=Max]

Outcome

[Resolved, Resolving, Not resolved, , applicable Terms of Use Resolved with sequelae, Death (from the event), Unknown]

Analytical methods:

For the above analysis item, the following analysis will be performed for each stratum of stratification factors.

- 1. Number of patients with ADRs
- 2. Number of ADRs
- 3. Percentage of patients with ADRs
- 4. Type of ADRs

All analyses will be accounted for as follows.

[Number of patients with ADRs]

Number of patients who experienced ADRs.

#### [Number of ADRs]

Number of ADRs When the same patient experienced multiple episodes of the same ADR, all episodes will be counted.

[Percentage of patients with ADRs]

Calculated as "Number of patients with ADRs/Number of patients in the safety analysis population x 100"

#### [Type of ADRs]

- ADRs will be coded using MedDRA/J. Events will be classified by SOC and then tabulated by PT. If the SOC is "Investigations", events will be sorted by HLGT (in ascending order of HLGT code, without output) and then tabulated by PT.
- Property of Takedai. For nonico The SOCs will be listed in the internationally agreed order for presentation of the number and percentage of patients with ADRs. When the same patient experienced multiple episodes of the same SOC, they will be counted only once for the SOC. For counting by category, episodes in the same SOC will be counted only once in the category of highest priority specified at the end of this section.
  - The PTs will be listed in ascending order of PT code for presentation of the number and percentage of patients with ADRs. When the same patient experienced multiple episodes of the same PT, they will be counted only once for the PT. For counting by category, episodes in the same PT will be counted only once in the category of highest priority as shown below.

Seriousness: Serious → Non-serious

25

Time to onset:  $1-27 \text{ days} \rightarrow 28-55 \text{ days} \rightarrow 56-83 \text{ days} \rightarrow 84-167$  $days \rightarrow 168-251 days \rightarrow 252-365 days \rightarrow 366 days or more$ 

# Analysis set: Safety analysis population Analysis item(s): ADRs Street: Analysis of the safety Analysis item(s): ADRs

[Male, Female] Stratification factors: Sex

Age (years)

[0<=-<5, 5<= -<10, 10<= -<15, Duration of Parkinson's disease

(years)

Inpatient/outpatient status (at [Outpatient, Inpatient]

initiation of treatment with this

drug)

Concurrent diseases [No, Yes]

Specific concurrent diseases

(patients counted under all [Diabetes mellitus, Hypertension,

applicable categories) Dyslipidemia, Hyperuricaemia]

Lifestyle-related disease [Hepatic steatosis, Alcoholic

hepatitis, Chronic hepatitis,

Hepatic disease Hepatic cirrhosis]

[Nephrotic syndrome,

Renal disease Glomerulonephritis, Chronic

renal failure]

Other diseases [Dementia, Pneumonia aspiration,

Constipation]

Dementia [No, Yes]

Property of Lakeda. For hopicolis Height (cm) [Min<= - <=140, 141<= - <=150,

151<= - <=160, 161<= - <=170,

 $171 \le - \le Max$ 

Min <= -<50, 50 <= -<65, 65 <= -Body weight (kg)

 $\leq = Max$ 

Smoking history [Never smoker, Current smoker, Former smoker, Unknown]

Modified Hoehn & Yahr Severity [0, 1, 1.5, 2, 2.5, 3, 4, 5]

scale (Stage)

Levodopa use at initiation of [No, Yes]

treatment with this drug

Wearing-off phenomenon [No, Yes]

Note: Only in patients given

levodopa at initiation of treatment

with this drug

Dyskinesia [No, Yes]

Note: Only in patients given

levodopa at initiation of treatment

with this drug

Concurrent renal disorder No, Yesl Concurrent hepatic disorder

Daily dose [1 mg, 0.5 mg, Other]

Overdose [No, Yes]

Note: Only when the daily dose was

"Other"

Any adverse event due to overdose [No, Yes]

Note: Only when overdose was

present

Reason for use (at initial dose)

Property of Takedai. For non-c' Note: Only when the daily dose was

"0.5 mg" or "Other"

[Because of the patient's mild hepatic impairment, low body weight, advanced age, or

concurrent CYP1A2 inhibitor use;

Other]

[AZILECT alone; AZILECT + Treatment stage

other Parkinson's disease

medication; Combined with only levodopa, without wearing-off phenomenon; Combined with levodopa and other Parkinson's disease medication, without

wearing-off phenomenon;

27

Combined with levodopa, with

wearing-off phenomenon]

Number of concomitant drugs [0 (AZILECT alone), 1 (AZILECT

+ another drug), ≥2 (AZILECT +

≥2 other drugs)]

Analytical methods: For the above analysis item, the following analysis will be performed for

each stratum of stratification factors.

1. Number of patients with ADRs

2. Percentage of patients with ADRs

All analyses will be accounted for as follows.

[Number of patients with ADRs]

• Number of patients who experienced ADRs.

[Percentage of patients with ADRs]

Calculated as "Number of patients with ADRs/Number of patients in the

safety analysis population x 100"

#### 4.4.2 Incidence of adverse drug reactions/infections by sex

Analysis set: Safety analysis population

Analysis item(s): ADRs

Stratification factors: Sex [Male, Female]

Analytical methods: The above item will be analyzed for each stratum of stratification factors

in a similar manner to Section 4.1.2.

#### 4.4.3 Incidence of adverse drug reactions/infections by age category (1)

Analysis set: Safety analysis population

Analysis item(s): ADRs

Stratification factors: Age (years)  $[Min \le -.65, 65 \le -.75, 75 \le -.75]$ 

<=Max

Analytical methods: The above item will be analyzed for each stratum of stratification factors

in a similar manner to Section 4.1.2.

#### 4.4.4 Incidence of adverse drug reactions/infections by age category (2)

Analysis set: Safety analysis population

Analysis item(s): ADRs relevant to the important identified risks in the safety specification

(i.e., Orthostatic hypotension, Somnolence and sudden onset of sleep,

Psychiatric symptoms such as hallucinations, Dyskinesia)

, 1 (AZILECT

≥2 (AZILECT +

gs)]

.g, 0.5 mg, Other]

[Min<= - <50, 50<= - <65, 65 ←

ymptoms <=Max]

Dyskinesia)
tementia [No, Yes]
ch as

resia [No, Yes] Stratification factor 1: Number of concomitant medications [0 (AZILECT alone), 1 (AZILECT (Orthostatic hypotension,

Psychiatric symptoms such as

hallucination)

Daily dose (Orthostatic

hypotension, Psychiatric symptoms such as hallucinations, Dyskinesia)

Body weight (kg) (Orthostatic

hypotension, Psychiatric symptoms such as hallucination, Dyskinesia)

Presence or absence of dementia

(Psychiatric symptoms such as

Presence or absence of dyskinesia

(Dyskinesia)

hallucinations)

Note: Only in patients given

levodopa at initiation of treatment

with this drug

Presence or absence of Wearing-off [No, Yes]

phenomenon (Orthostatic

hypotension, Psychiatric symptoms

such as hallucination)

Note: Only in patients given

levodopa at initiation of treatment

with this drug

Duration of Parkinson's disease  $[0 \le - <5, 5 \le - <10, 10 \le - <15,$ 

(years) (Orthostatic hypotension,  $15 \le - \le Max$ 

Psychiatric symptoms such as

hallucination)

Stratification factor 2: [Min<= - <65, 65<= - <75, 75<= -Age (years)

 $\leq Max$ 

Analytical methods: The above analysis item by risk item will be analyzed as follows, with stratification by Stratification factor 1 and Stratification factor 2. For the

risk items to be analyzed, the definitions described in the safety specification (important identified risks, important potential risks, and

important missing information) shall be followed.

1. Number of patients with ADRs

#### 2. Percentage of patients with ADRs

#### 4.4.5 Incidence of adverse drug reactions/infections by duration of Parkinson's disease

Safety analysis population Analysis set:

**ADRs** Analysis item(s):

[0<= - <5, 5<= - <10, 10<= - <15, 15<= - <=Max] Stratification factors: Duration of Parkinson's disease

(years)

Analytical methods: The above item will be analyzed for each stratum of stratification factors

in a similar manner to Section 4.1.2.

#### 4.4.6 Incidence of adverse drug reactions/infections by presence or absence of concurrent diseases

Safety analysis population Analysis set:

Analysis item(s): **ADRs** 

Stratification factors: Concurrent diseases

The above item will be analyzed for each stratum of stratification factors Analytical methods:

in a similar manner to Section 4.1.2.

#### 4.4.7 Incidence of adverse drug reactions/infections by body weight

Analysis set: Safety analysis population

Analysis item(s):

[Min<= - <50, 50<= - <65, 65<= -Stratification factors: Body weight (kg)

The above item will be analyzed for each stratum of stratification factors Analytical methods:

in a similar manner to Section 4.1.2.

#### 4.4.8 Incidence of adverse drug reactions/infections by presence or absence of concurrent renal disorder

Analysis set: Safety analysis population

Analysis item(s): **ADRs** 

Stratification factors: Concurrent renal disorder [No, Yes]

Analytical methods: The above item will be analyzed for each stratum of stratification factors

in a similar manner to Section 4.1.2.

#### 4.4.9 Incidence of adverse drug reactions/infections by presence or absence of concurrent hepatic disorder

Analysis set: Safety analysis population Analysis item(s): ADRs

Stratification factors: Concurrent hepatic disorder [No, Yes]

Analytical methods: The above item will be analyzed for each stratum of stratification factors

in a similar manner to Section 4.1.2.

#### 4.4.10 Incidence of adverse drug reactions/infections by treatment stage

Analysis set: Safety analysis population

Analysis item(s): ADRs

Stratification factors: Treatment [AZILECT alone; AZILECT + other Parkinson's disease

stage medication; Combined with only levodopa, without

wearing-off phenomenon; Combined with levodopa and other Parkinson's disease medication, without wearingoff phenomenon; Combined with levodopa, with

wearing-off phenomenon]

Analytical methods: The above item will be analyzed for each stratum of stratification factors

in a similar manner to Section 4.1.2.

#### 4.4.11 Incidence of adverse drug reactions/infections by daily dose

Analysis set: Safety analysis population

Analysis item(s): ADRs

Stratification factors: Daily dose [1 mg, 0.5 mg, Other]

Analytical methods: The above item will be analyzed for each stratum of stratification factors

in a similar manner to Section 4.1.2.

#### 4.4.12 Incidence of adverse drug reactions/infections by presence or absence of dementia

Analysis set: Safety analysis population

Analysis item(s): ADRs

Stratification factors: Dementia [No, Yes]

Analytical methods: The above item will be analyzed for each stratum of stratification factors

in a similar manner to Section 4.1.2.

#### 4.4.13 Incidence of adverse drug reactions/infections by presence or absence of dyskinesia

Analysis set: Safety analysis population

Analysis item(s): ADRs

Stratification factors: Dyskinesia [No, Yes]

Note: Only in patients given

Properly of Takeda: For non-commercial use only and subject to the applicable Tames of Use

#### 5 Efficacy data

#### 5.1 UPDRS Part III total score over time

Analysis set: Efficacy analysis population
Analysis item(s): UPDRS Part III total score

Time point of Baseline, 6 months, 12 months, 18 months, and 24 months of treatment or

assessment: discontinuation, final assessment

Analytical methods: For the above analysis item, summary statistics at each time point of

assessment will be presented for the measured value and change (Postbaseline score at respective time point – Baseline score). A line graph will

be created for the change.

#### 5.2 UPDRS Part III tremor score over time

Analysis set: Efficacy analysis population
Analysis item(s): UPDRS Part III tremor score
Time point of Baseline, final assessment

assessment:

Analytical methods: For the above analysis item, summary statistics at each time point of

assessment will be presented for the measured value and change (Score at

final assessment - Baseline score).

#### 5.3 UPDRS Part III akinesia/hypokinesia score over time

Analysis set: Efficacy analysis population

Analysis item(s): UPDRS Part III akinesia/hypokinesia score

Time point of Baseline, final assessment

assessment:

Analytical methods: For the above analysis item, summary statistics at each time point of

assessment will be presented for the measured value and change (Score at

final assessment - Baseline score).

#### 5.4 UPDRS Part III rigidity score over time

Analysis set: Efficacy analysis population
Analysis item(s): UPDRS Part III rigidity score
Time point of Baseline, final assessment

assessment:

Analytical methods: For the above analysis item, summary statistics at each time point of

assessment will be presented for the measured value and change (Score at

final assessment – Baseline score).

#### 5.5 Factors likely affecting the efficacy

#### 5.5.1 Factors likely affecting the efficacy

Analysis set: Efficacy analysis population UPDRS Part III total score Analysis item(s):

At 6 months, 12 months, 18 months, and 24 months of treatment with this Time point of

drug or discontinuation, final assessment assessment:

Stratification factors: Duration of Parkinson's disease [0<= - <5, 5<= - <10, 10<= - <15,

(years)

Body weight (kg)

<=Max]

[0, 1, 1.5, 2, 2.5, 3, 4, 5] Modified Hoehn & Yahr Severity

scale (Stage)

Any drugs to treat Parkinson's [No, Yes]

disease other than AZILECT and

levodopa

Number of concomitant drugs [0 (AZILECT alone), 1 (AZILECT

+ another drug), ≥2 (AZILECT +

 $\geq 2$  other drugs)]

Treatment stage

Treatment stage [AZILECT alone; AZILECT +

other Parkinson's disease

medication; Combined with only levodopa, without wearing-off phenomenon; Combined with levodopa and other Parkinson's disease medication, without wearing-off phenomenon; Combined with levodopa, with wearing-off phenomenon]

[Min<= - <65, 65<= - <70, 70<= -

<75, 75 <= - <80, 80 <= - <= Max

Analytical methods: For the above analysis item, for each stratum of stratification factors,

summary statistics of the change (Post-baseline score at respective time point – Baseline score) at each time point of assessment will be presented.

#### 5.5.2 UPDRS Part III total score by age category and number of concomitant drugs

Analysis set: Efficacy analysis population
Analysis item(s): UPDRS Part III total score

Time point of Baseline, 12 months, and 24 months of treatment or discontinuation, final

assessment: assessment

Stratification factor 1: Number of [0 (AZILECT alone), 1 (AZILECT + another drug),

concomitant drugs  $\geq 2$  (AZILECT +  $\geq 2$  other drugs)]

Stratification factor 2: Age (years)  $[Min \le -.. < 65, 65 \le -.. < 70, 70 \le -.. < 75, 75 \le -.. < 80,$ 

 $80 \le - \le Max$ 

Analytical methods: For the above analysis items, with stratification by Stratification factor 1

and Stratification factor 2, summary statistics of the change at each time

point of assessment (Post-baseline score at respective time point –

Baseline score) will be presented.

## 5.5.3 Number of patients continuing treatment with this drug by age category and number of concomitant drugs

Analysis set: Efficacy analysis population

Analysis item(s): Patients who continue to receive this medication

Time point of At 6 months and 12 months of treatment with this drug

assessment:

Stratification factor 1: Number of [0 (AZILECT alone), 1 (AZILECT + another drug),

concomitant drugs  $\geq 2$  (AZILECT +  $\geq 2$  other drugs)]

Stratification factor 2: Age (years) [Min<= - <65, 65<= - <70, 70<= - <75, 75<= - <80,

 $80 \le - \le Max$ 

Analytical methods: For the above analysis item, with stratification by Stratification factor 1

and Stratification factor 2, the discrete data at each time point of

assessment will be summarized using frequency tabulation.

#### 5.5.4 Number of patients continuing treatment with this drug by age category

Analysis set: Efficacy analysis population

Analysis item(s): Patients who continue to receive this medication

Time point of At 6 months and 12 months of treatment with this drug

assessment:

Stratification factors:

Daily dose [1 mg, 0.5 mg]

Tor the above analysis item, for each squency tabular. Analytical methods:

#### 5.5.5 Number of patients continuing treatment with this drug by dose

Analysis set:

Analysis item(s):

Time point of

assessment:

Stratification factors:

Property of Takeda. For non-commercial use only and parties of the property of Takeda. Analytical methods:

#### Incidence of adverse drug reactions/infections in the additional pharmacovigilance plan

# Incidence of adverse drug reactions/infections in the additional pharmacovigilance plan 6.1 The above analysis item will be analyzed for each stratum of stratification factors, in accordance with Re-examination Notification No. 0325-10 accordance with Re-examination No. 0325-10 (Attached Form 12)

Analysis set:

Analysis item(s):

Stratification

factors:

Analytical

methods:

For the risk names and the listing order of the risk names, the definitions Property of Takeda. For non-commercial use only and described in the safety specification (important identified risks, important potential risks, and important missing information) shall be followed.

#### Summary of patients in the post-marketing survey/study

#### Summary of patients in the post-marketing survey/study (Attached Form 16) 7.1

Safety analysis population Analysis set:

Analysis item(s): Patient ID number

Name of medical institution

Sex

Date of birth

Reason for use (disease code, disease name)

Concurrent disease (disease code, disease name)

Route of administration

Maximum dose

Average dose

Units

Therapy dates (AZILECT therapy period)

Concomitant drug (drug code, drug name)

Degree of effect

Adverse drug reaction (disease code, disease name, outcome)

CRF No.

Dropout

Reason for dropout

Adverse drug reaction (safety specification, fall or trauma, accident or trauma)

For the above analysis item, a tabulated list will be prepared in accordance with Analytical

the rules for data entry and file preparation stipulated by Re-examination methods:

Phan 2020. Notification No. 1119-3 of the Pharmaceutical Evaluation Division,

Pharmaceutical Safety and Environmental Health Bureau, dated November 19,

#### **History of this document (Version control)**

| Version | Date | Prepared/revised by | Comments | |
|---|---|---|---|---|
| Initial<br>version | 2022.4.15 | PPD | Preparation of initial version | ermsoft |

Property of Takeda: For noncommercial use only and subject to the applicable Test